CLINICAL TRIAL: NCT04186858
Title: Assessment of Levels of Intracellular Cytokines and Markers in Cells Recovered From the Anterior Eye (Phase 4)
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-6316
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Impression Cytology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ocular surface cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic: Based on the score of the questionnaire, eligible subjects will be placed in the Symptomatic group where cell samples will be collected from the front surface of the subject's eyes.
- Asymptomatic: Based on the score of the questionnaire, eligible subjects will be placed in the Asymptomatic group where cell samples will be collected from the front surface of the subject's eyes.

SUMMARY:
This is a single-visit, non-randomized, bilateral, cross-sectional study. In a pre-screening assessment, potential subjects will be invited to complete a web-based questionnaire that is validated to determine symptomatic vs asymptomatic contact lens wearers. Results of this questionnaire will be used to determine whether subjects are eligible to proceed to Visit 1. During Visit 1, cell samples will be collected from the front surface of the subject's eyes.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 45 years of age (inclusive) at the time of screening
  4. They have worn the same brand of soft contact lenses for at least the previous three months.
  5. They agree not to participate in other clinical research trials for the duration of this study.
  6. In a pre-study screening assessment, they must have a CLDEQ-8 score of 10 or less (asymptomatic group) or 20 or higher (symptomatic group).
  7. They possess a wearable pair of distance glasses and agree to bring these to the study visit (if needed for distance vision correction).
  8. They can attain a high contrast logMAR visual acuity of 0.20 or better in their habitual contact lenses.
  9. Their habitual contact lenses fit satisfactorily.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study
  3. They have an ocular disorder which would normally contraindicate contact lens wear.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  7. They have taken part in any other contact lens or care solution clinical trial research, within two weeks prior to starting this study.
  8. They are regularly (once per day or more) using oral or inhaled steroids or anti-inflammatory medications.
  9. They are using any topical medications such as eye drops or ointments.
  10. History of allergic reaction to sodium fluorescein or topical anesthetic.
  11. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  13. They have Grade 3 or greater of any of the following ocular surface signs: corneal edema, corneal vascularization, corneal staining (white light evaluation), tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
  14. Any active ocular infection or inflammation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible subjects aged 18 years and above with normal healthy eyes will be recruited for this work.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Number of Cells | ~6 hours of contact lens wear time
  The frequency count of cells will be summarized within the category
Types of Cells | ~6 hours of contact lens wear time
  The percentage of types of cells will be summarized within the category.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu